CLINICAL TRIAL: NCT05500196
Title: Impact of Gastric Length of Myotomy During Poem on Gastroesophageal Reflux : A Randomized Controlled Trial
Brief Title: Impact of Gastric Length of Myotomy During POEM on Gastroesophageal Reflux
Acronym: IGL
Status: Completed | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, PRINCIPAL INVESTIGATOR, Asian Institute of Gastroenterology, India
Other Study IDs: POEM 005
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Gastric Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myotomy length: Extended myotomy >2.5cm
  Interventions: Device: Per Oral Endoscopy Myotomy (POEM)
- MYOTOMY LENGTH: Extended myotomy>3
  Interventions: Device: Per Oral Endoscopy Myotomy (POEM)

INTERVENTIONS:
Device: Per Oral Endoscopy Myotomy (POEM) — POEM is a form of natural orifice transluminal endoscopic surgery that is completed by creating a submucosal tunnel in the lower part of esophagus to reach the inner circular muscle bundles of the LES to perform myotomy, while preserving the outer longitudinal muscle bundles. The result is decreased resting pressure of the LES, facilitating the passage of ingested material.

SUMMARY:
This observational study will be conducted among 43 patients of both sexes in each group Study participants will be of the age more than 18 years

* STUDY PROCEDURE-Pre-defined technique to avoid bias and confounding due to multiple factors
* All the poem procedures will be performed by posterior route
* Preservation of sling fibers will be attempted in all the cases to avoid heterogeneity
* Length of esophageal myotomy will be kept constant (4-6cm)
* Double scope technique will be utilized to confirm the gastric extent of myotomy

First evaluation at 1-month: based on Symptoms

• Second evaluation: at 6 months by

* Objective evaluation: UGI endoscopy, High resolution manometry, Timed barium swallow
* Eckardt score, GERD-HRQL
* 24-hour pH study with manual readings

DETAILED DESCRIPTION:
• The primary outcome of the study is the incidence of significant reflux esophagitis (≥grade B) in cases with standard and extended gastric myotomies at 6 months after POEM

Secondary outcomes:

* Significant esophageal acid exposure (>6%) as defined by the revised Lyon consensus
* Symptoms of GERD (GERD HRQL)
* Clinical efficacy (Eckardt score≤3)
* Esophageal emptying at 5 minutes
* High resolution manometry parameters (LES pressures and Integrated relaxation pressure in mmhg units)
* All the secondary outcomes will be assessed at 6 months after poem procedure

Eligibility:

Eligible cases with idiopathic achalasia (type I and II) will be enrolled in the study and randomized (1:1 ratio) in two groups according to the length of gastric myotomies

INCLUSION CRITERIA :

* Idiopathic achalasia (type I and II)
* Age ≥18 years
* Willing to provide informed consent and comply with the study protocol

Exclusion criteria

* Ineligibility for POEM procedure
* Spastic esophageal motility disorders
* Presence of esophageal diverticulum and hiatal hernia
* Prior hellers myotomy with or with out fundoplication

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic achalasia (type I and II)
* Age ≥18 years
* Willing to provide informed consent and comply with the study protocol

Exclusion Criteria:

* Ineligibility for POEM procedure
* Spastic esophageal motility disorders
* Presence of esophageal diverticulum and hiatal hernia
* Prior hellers myotomy with or with out fundoplication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible cases with idiopathic achalasia(type I & II) will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Impact of Gastric Length of myotomy during poem on Gastroesophageal reflux | 6 months
  incidence of reflux esophagitis >grade B in cases with standard and extended gastric myotomies after POEM
Ph metry test for gastroesophageal reflux | 6 months
  Significant esophageal acid exposure(> 6%)

SECONDARY OUTCOMES:
Symptoms of Gastro esophageal reflux disease | 6 months
  Health related quality of life questionaires or scores in numericals
High resolution manometry parameters(LES pressures and IRP) | 6 months
  lower esophageal sphincter pressure will be assesed by mmhg, integrated resting pressure in mmhg units

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Nabi, MBBS MD DNB, Study Director — ASIAN INSTITUTE OF GASTROENTEROLOGY/AIG HOSPITALS
Locations (1):
- Asian Institute of Gastroenterology /Aig Hospitals, Hyderabad, Telangana, India